CLINICAL TRIAL: NCT01097395
Title: Concentration-Controlled Ribavirin for the Treatment of Patients With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-1198; K23DK082621 (NIH)
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis C Virus
Keywords: ribavirin; pharmacokinetics; Hepatitis C virus
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Weight-Based Ribavirin Dosing (Active Comparator): 1000 mg daily in patients weighing <75 kg and 1200 mg daily in patients weighing ≥ 75 kg
  Interventions: Drug: ribavirin
- Concentration-Controlled Ribavirin Dosing (Experimental): Dose adjusted based on first dose AUC0-12
  Interventions: Drug: ribavirin

INTERVENTIONS:
Drug: ribavirin — Randomization to standard weight based ribavirin dosing (1000 or 1200 mg daily) or concentration-guided dosing based on first dose AUC0-12

SUMMARY:
The purpose of this study is to determine if concentration-controlled ribavirin dosing can achieve a targeted level of plasma exposures and if it appears safe and effective compared with standard weight-based ribavirin dosing. Forty, previously treatment-naive participants with genotype 1 disease will be randomized to receive concentration-guided or standard weight-based ribavirin. Peginterferon alfa 2a,ribavirin, and telaprevir will be provided through the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV-infected men and women
* 18-70 years
* HCV genotype 1
* Deemed ready for HCV treatment by hepatology provider and patient
* Allowed medications: all those not specifically listed in the exclusion criteria below including medications for peginterferon / ribavirin - related adverse effects: acetaminophen, ibuprofen, diphenhydramine, selective serotonin reuptake inhibitors, darbepoeitin, erythropoietin, GCSF

Exclusion Criteria:

* previous treatment with interferon, peginterferon, investigational HCV drugs, boceprevir, or ribavirin;
* baseline absolute neutrophil count (ANC) < 1000/mm3,
* platelets < 100,000/mm3,
* hemoglobin < 12 g/dL for women and < 13 g/dL for men;
* HIV positive serostatus;
* HBV positive serostatus;
* decompensated liver disease (i.e., ascites, history of esophageal variceal bleeding, hepatic encephalopathy);
* autoimmune hepatitis
* hemoglobinopathy (e.g., sickle cell anemia, thalassemia)
* Cockcroft and Gault estimated creatinine clearance < 50 mL/min;
* alcohol or illicit drug use that in the opinion of the investigator would interfere with study participation and/or impact study results
* for females, active pregnancy or any intent to become pregnant during study period or for up to 6 months after completing treatment
* for males, a pregnant female partner or intent to impregnate a female during study period or for up to 6 months after completing treatment
* for both sexes an unwillingness to use two forms of contraception during the study period and for 6 months after completing treatment. While on telaprevir and for 2 weeks following discontinuation of telaprevir, females must use two non-hormonal forms of contraception;
* history of significant or unstable cardiac disease including severe coronary artery disease (unstable angina, recent myocardial infarction, chest pain with exertion) or congestive heart failure;
* receipt of an organ transplant;
* malignant neoplastic disease;
* chronic pulmonary disease that in the opinion of the study hepatologists would preclude treatment with peginterferon and ribavirin (e.g., pulmonary function tests ≤70% within the previous 2 years);
* history of admission to a psychiatric facility within the previous year;
* suicide attempt within the previous 3 years;
* concomitant medications including: amantadine, mycophenolate mofetil, and investigational HCV compounds, alfuzosin, alfentanil, ergot derivatives (dihydroergotamine/ergotamine/ergonovine/methylergonovine), meperidine, anti-arrhythmics (quinidine, flecainide, propafenone, amiodarone, bepridil), astemizole, terfenadine, buspirone, diazepam, estazolam, oral midazolam, triazolam, budesonide, domperidone, eletriptan, eplerenone, fluticasone, pimozide, salmeterol, calcium channel blockers (diltiazem, felodipine, nifedipine, nisoldipine, verapamil), cisapride, cyclosporine, sirolimus, systemic tacrolimus, atorvastatin, lovastatin, simvistatin, sildenafil, tadalafil, verdenafil, antibiotics (clarithromycin, erythromycin, telithromycin, troleandomycin), carbamazepine, Phenobarbital, phenytoin, nefazodone, St. Johns Wort, antifungals (fluconazole, itraconazole, ketoconazole, posaconazole, voriconazole), rifampin, rifabutin, aprepitant, cholestyramine, fluvoxamine, mifepreistone, modafinil, systemic dexamethasone. With the exception of St. Johns Wort, investigators may use their discretion on use of herbal and dietary supplements.
* Evidence of severe retinopathy or clinically relevant ophthalmologic disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Kiser, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Wu LS, Rower JE, Burton JR Jr, Anderson PL, Hammond KP, Baouchi-Mokrane F, Everson GT, Urban TJ, D'Argenio DZ, Kiser JJ. Population pharmacokinetic modeling of plasma and intracellular ribavirin concentrations in patients with chronic hepatitis C virus infection. Antimicrob Agents Chemother. 2015 Apr;59(4):2179-88. doi: 10.1128/AAC.04618-14. Epub 2015 Feb 2. PMID 25645847

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Weight-Based Ribavirin Dosing | Concentration-Controlled Ribavirin Dosing
Started | 17 | 18
Completed | 14 | 14
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Weight-Based Ribavirin Dosing | Concentration-Controlled Ribavirin Dosing | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (10.2) | 53.4 (5.9) | 50.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 15 | 15 | 30
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Ribavirin AUC-12 Variability
Description: Demonstrate that concentration-controlled ribavirin dosing can achieve a targeted level of plasma exposure with reduced variability in the steady-state area-under-the-concentration-time curve (AUC0-12) compared with standard weight-based ribavirin dosing
Time Frame: steady state (~weeks 9-10)
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Standard Weight-Based Ribavirin Dosing | Concentration-Controlled Ribavirin Dosing
Number analyzed (Participants) | 17 | 18
ng*hr/mL | 34425 (10046) | 40903 (10953)

2. Secondary Outcome: Safety - Absolute Hemoglobin Declines
Time Frame: from baseline through end of treatment, up to 48 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Standard Weight-Based Ribavirin Dosing | Concentration-Controlled Ribavirin Dosing
Number analyzed (Participants) | 17 | 18
g/dL | 2.6 (1.9) | 3.6 (1.2)

3. Secondary Outcome: Sustained Virologic Response (i.e., Cure)
Description: Compare proportions with SVR in standard weight-based vs. concentration-guided ribavirin dosing groups. Number of participants with sustained virologic response is reported.
Time Frame: assessed 12 weeks after stopping treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Weight-Based Ribavirin Dosing | Concentration-Controlled Ribavirin Dosing
Number analyzed (Participants) | 17 | 18
Participants | 8 | 12

ADVERSE EVENTS:
Time Frame: 48 Weeks
Arm/Group | Standard Weight-Based Ribavirin Dosing | Concentration-Controlled Ribavirin Dosing
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 4/17 | 7/18
Other Adverse Events (participants affected / at risk) | 14/17 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Weight-Based Ribavirin Dosing (N=17) | Concentration-Controlled Ribavirin Dosing (N=18)
Hemoglobin < 8.5 g/dL (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Chest pain (Cardiac disorders) | 1 (1) | 1 (1)
Frozen arms (Nervous system disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tooth pain and vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mood alteration (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Weight-Based Ribavirin Dosing (N=17) | Concentration-Controlled Ribavirin Dosing (N=18)
Hemoglobin < 10 g/dL (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
ANC < 1000/mm3 (Blood and lymphatic system disorders) | 9 (9) | 5 (5)
Platelets < 75,000/mm3 (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
WBC <2000/mm3 (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Grade 3 Depression (Nervous system disorders) | 1 (1) | 1 (1)
Grade 3 Fatigue (Nervous system disorders) | 2 (2) | 1 (1)
Grade 3 Insomnia (Nervous system disorders) | 2 (2) | 0 (0)
Grade 3 Mood Alteration (Nervous system disorders) | 2 (2) | 0 (0)
Grade 3 Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Grade 3 Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No